CLINICAL TRIAL: NCT04507516
Title: A Pilot Study on the Effects of Medically Supervised, Water-Only Fasting and Refeeding on Cardiometabolic Risk
Brief Title: Fasting for Brain and Heart Health (FBHH)
Acronym: FBHH
Status: Completed | Type: Observational
Sponsor: TrueNorth Health Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TNHF2018-1
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, sera
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Water-only Fasting Cohort: Obese/overweight, non-diabetic patients undergoing elective water-only fasting treatment.
  Interventions: Other: Water-only Fasting

INTERVENTIONS:
Other: Water-only Fasting — Water-only fasting for at least 10 days followed by 5 days of refeed.

SUMMARY:
This pilot study is designed to investigate the effect of water-only fasting and refeeding on the homeostatic model of insulin resistance (HOMA-IR), a measure of insulin resistance.

DETAILED DESCRIPTION:
Ischemic stroke is a leading cause of death and a major public health burden. Data suggests that insulin resistance is a potential risk factor for cardiovascular disease, including ischemic stroke, and that dietary and lifestyle intervention can reduce insulin resistance as well as these disease risks. Nonetheless, current intervention strategies have done little to reduce overall stroke incidence. Therefore, an intervention, such as prolonged medically supervised water-only fasting, might be an effective strategy to both reduce insulin resistance and encourage dietary and lifestyle changes that reduce incidence of stroke.

This pilot study is designed to investigate the effect of water-only fasting and refeeding on the homeostatic model of insulin resistance (HOMA-IR), a measure of insulin resistance. Additionally, the study will assess if markers of cardiovascular health and inflammation change before and after water-only fasting. Water-only fasting participants will be recruited from patients who voluntarily elect to water-only fast for 10 or more consecutive days. Clinical variables and blood will be collected at baseline, every 7th day during fasting and refeeding, and the final day of fasting and refeeding.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* 40-70 years old
* Fasting plasma glucose <12 6mg/dL and/or hemoglobin A1c <7%
* Body Mass Index (BMI) >25 kg/m2
* Elect and qualify for a water-only fast of at least 10 consecutive days
* Provide informed consent

Exclusion Criteria:

* Active malignancy
* Active inflammatory disorder including classic autoimmune connective tissue (Lupus, Sjogrens, ANCA), multiple sclerosis, and inflammatory bowel disorders (Ulcerative colitis, Crohn's)
* Stroke or heart attack within the last 90 days

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Overweight and obese, non-diabetic participants recruited from voluntary patients.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Changes in insulin resistance from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  Insulin resistance assessed using serum glucose and insulin to calculate homeostatic model of insulin resistance (HOMA-IR) [fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5]

SECONDARY OUTCOMES:
Changes in lipid profile from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  Lipid profile assessed using serum to measure cholesterol, triglycerides, high-density lipoprotein (HDL), and low-density lipoprotein (LDL) and reported in mg/dL
Changes in weight from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  Weight measured on a digital scale and reported in kilograms (kg)
Changes in resting systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  SBP and DBP measured using digital blood pressure device and reported in mmHg
Changes in abdominal circumference from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  Abdominal circumference measured on bare skin at the minimal waistline with a tension-sensitive, non-elastic tape and reported in centimeters (cm)
Changes in high sensitivity C-reactive protein (hsCRP) from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast
  hsCRP assessed using serum and reported in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Toshia R Myers, PhD, Principal Investigator — Director
Locations (1):
- TrueNorth Health Center, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: Undecided